CLINICAL TRIAL: NCT05458830
Title: Breaking Down Barriers to a Suicide Prevention Helpline: a Web-based Randomised Controlled Trial
Brief Title: Breaking Down Barriers to a Suicide Prevention Helpline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 113 Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Selftest113; 2021.0443 (Other: Medical Ethics Committee VUMC)
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-07

CONDITIONS: Suicidal Ideation
Keywords: Barrier reduction intervention; Suicidal ideation; Self-help; Suicide prevention helpline; Randomised controlled trial; Help-seeking
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomised controlled trial for the anonymous users of an online self-test for suicidal thoughts in which individuals with severe suicidal thoughts and no interest in contacting the helpline will be randomly allocated either to a short barrier reduction intervention (BRI) or receive a general advisory text (care as usual). To minimise the burden on the high-risk and sensitive study population, the investigators aim that it is feasible to complete the intervention within 10 minutes.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After selecting a barrier in the barrier survey, participants receive tailored information with the purpose of addressing common concerns and misconceptions about the helpline.
  Interventions: Behavioral: Brief Barrier Reduction Intervention
- Care as usual (Other): Plain advisory text
  Interventions: Behavioral: Plain advisory text

INTERVENTIONS:
Behavioral: Brief Barrier Reduction Intervention — After selecting a barrier in the barrier survey, participants receive tailored information with the purpose of addressing common concerns and misconceptions about the helpline.
  Arms: Intervention
Behavioral: Plain advisory text — Care as usual
  Other Names: care as usual
  Arms: Care as usual

SUMMARY:
Every month, around four thousand people fill in the anonymous self-test for suicidal thoughts on the website of the Dutch suicide prevention helpline 113 Suicide Prevention. The self-test includes the Suicidal Ideation Attributes Scale (SIDAS) and informs people about the severity of their suicidal thoughts. The vast majority (70%) of people who complete the test score higher than the cut-off point (≥ 21) for severe suicidal thoughts. Despite this, only around 10% of test-takers navigate to the webpage about contacting the helpline.

In this study the investigators test an intervention that aims to reduce barriers to contacting the helpline via chat or phone. People with severe suicidal thoughts and little motivation to contact the helpline will be randomly allocated either to a brief Barrier Reduction Intervention (BRI) or care as usual, a plain advisory text.

The aim of our study is two-fold: (i) to measure the effectiveness of a brief barrier reduction intervention (BRI) in the self-test motivating people with severe suicidal thoughts to contact the helpline, and (ii) to specifically evaluate the effectiveness of the intervention in increasing service utilisation by high-risk groups for suicide such as men and people of middle age.

DETAILED DESCRIPTION:
Research suggests that people with suicidal thoughts often do not seek help, making them invisible for preventive measures and targeted support. Anonymous online help can be a low-threshold first step towards professional face-to-face help. In the Netherlands, the suicide prevention organisation '113 Suicide Prevention' provides around-the-clock anonymous support by phone and chat, as well as an online self-help course, self-assessment tests and brief online coaching and therapy. Apart from the homepage, the 'test yourself' page is the most visited section of the helpline's website. Every month, more than 4,000 people fill in the anonymous self-test for suicidal thoughts. This self-test includes the Suicidal Ideation Attributes Scale (SIDAS) and informs the test-taker of the severity of their suicidal thoughts. Although the vast majority of people who complete the test score higher than the cut-off point for severe suicidal thoughts, only approximately 10% of test-takers go on to navigate to the web-page about contacting the helpline. And although due to the anonymity of the helpline's services it is not possible to know if people follow up the advice of contacting the helpline, the difference in demographic distributions between the users of the self-test and the crisis helpline confirms the assumption that a substantial group does not continue using helpline service. While the percentage of men among the self-test users is 40%, it is only around 25% among the users of the helpline.

The study is designed as a randomised controlled trial for the anonymous users of an online self-test for suicidal thoughts in which individuals with severe suicidal thoughts and no interest in contacting the helpline will be randomly allocated either to a short barrier reduction intervention (BRI) or receive a general advisory text (care as usual). To minimise the burden on our high-risk and sensitive study population, the investigators aim that it is feasible for the participants to complete the intervention within 10 minutes.

The aim of our study is two-fold: (i) to measure the effectiveness of a brief barrier reduction intervention (BRI) in the self-test motivating people with severe suicidal thoughts to contact the helpline, and (ii) to specifically evaluate the effectiveness of the intervention in increasing service utilisation by high-risk groups for suicide such as men and people of middle age.

ELIGIBILITY:
Exclusion Criteria:

* participant is younger than 16 years old.
* participant scores below the cut-off point for severe suicidal thoughts (SIDAS score < 21).
* participant scores above the cut-off point for severe suicidal thoughts (SIDAS score ≥ 21) and reports being likely to contact the suicide prevention helpline. They will be directly transferred to the contact details of the helpline.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
The use of a direct link to the helpline | immediately after intervention
  The primary outcome measure is the use of a direct link to the helpline after completing the intervention or the control condition (plain advisory text, care as usual).

SECONDARY OUTCOMES:
Self-reported likelihood of contacting the helpline | immediately after intervention
  Due to the anonymous nature of the helpline, it is not possible to measure if people who do not directly use the link to the helpline, contact the helpline at a later point in time. Therefore, the self-reported likelihood of contacting the helpline (5-point interval scale, ranging from not likely to very likely) is included as a proxy measurement.

OTHER OUTCOMES:
Severity of suicidal thoughts: Suicidal Ideation Attributes Scale (SIDAS) | Baseline measurement
  Score on the Suicidal Ideation Attributes Scale (SIDAS). The SIDAS consists of five items on a 10-point scale measuring the frequency of suicidal thoughts, controllability, closeness to attempt, distress and interference with daily activities. Total scores range from 0 to 50, with higher scores indicating more severe suicidal thoughts.
Gender | Baseline measurement
  Self-reported gender identity (male/female/other)
Age group | Baseline measurement
  Self-reported age group
Receiving treatment for mental health problems | Baseline measurement
  Currently receiving treatment for mental health problems (yes/no/on waiting list)
Satisfaction with the self-test | immediately after intervention
  Respondents' satisfaction with the self-test (intervention or control condition). 4 point-scale ranging from poor to excellent with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Mérelle, Principal Investigator — 113 Suicide Prevention
Locations (1):
- 113 Suicide Prevention, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data will be made available upon request

REFERENCES:
- [Derived] van der Burgt MCA, Merelle S, Brinkman WP, Beekman ATF, Gilissen R. Breaking Down Barriers to a Suicide Prevention Helpline: Protocol for a Web-Based Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 24;12:e41078. doi: 10.2196/41078. PMID 37093641